CLINICAL TRIAL: NCT05510947
Title: Acute Postoperative Pain and Catastrophizing in Patients Undergoing Unicompartmental Knee Arthroplasty - A Prospective, Observational, Single-center, Cohort Study
Brief Title: Acute Postoperative Pain and Catastrophizing in Patients Undergoing Unicompartmental Knee Arthroplasty
Acronym: KATUKA
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Deichmann Springborg, MD, PhD-student, Copenhagen University Hospital, Hvidovre
Other Study IDs: UKAPCS
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Post Operative Pain
Keywords: Acute Postoperative Pain; Unicompartmental Knee Arthroplasty; Pain catastrophizing scale
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Advantages of unicompartmental knee arthroplasty (UKA) compared to total knee arthroplasty (TKA) include shorter hospital stays, faster recovery, fewer infections and readmission, and lower costs. It is well documented in TKA-surgery that high pain responders (HPR), evaluated using the Pain Catastrophizing Scale (PCS), have higher postoperative pain responses compared to low pain responders (LPR). These HPR-patients constitute a vulnerable high risk patient group and potentially benefit from targeted treatment. Currently, the distribution of HPR- and LPR-patients and their association with acute pain following UKA is not well investigated. The knowledge that this research project generates is essential to determine how studies with analgesia interventions should be designed. In the future this will contribute in targeting treatment for high risk patient groups to reduce pain and improve postoperative mobilization, and ultimately decrease length of hospital stay in patients undergoing UKA. By targeting treatment, a potential overtreatment is also avoided.

The aim of this study is to investigate the prevalence of high- and low-pain responders, defined by a PCS score > 20 and ≤ 20 respectively, as well as the acute postoperative course of pain for these groups after unicompartmental knee arthroplasty.

DETAILED DESCRIPTION:
Background:

Primary knee arthroplasty is a frequently performed procedure and is expected to increase in numbers over the next decade. Advantages of unicompartmental knee arthroplasty (UKA) compared to total knee arthroplasty (TKA) include shorter hospital stays, faster recovery, fewer infections and readmissions, and lower costs. The length of hospital stay after UKA is variable, but an increased length of hospitalization has been associated with more complications and higher readmission rates. A recent study has shown that the main reasons for continued hospitalization beyond 24 hours after surgery are pain and lack of mobilization. Strategies to decrease the length of stay after UKA should thus be aimed at improved analgesia and postoperative mobilization.

There is a large interindividual variability in the postoperative pain response. It is well documented in TKA-surgery that high pain responders (HPR), evaluated using the Pain Catastrophizing Scale (PCS), have higher postoperative pain responses compared to low pain responders (LPR). Recently, it has been shown that HPR patients undergoing TKA benefit from a larger preoperative dose of glucocorticoid compared to a previously recommended dose. Interestingly, the same difference has not been found in LPR patients (Nielsen et al.: IN PREPARATION, clinicaltrials.gov ID NCT03758170, EudraCT 2018-002634-20, VEK H-18034756). These HPR patients constitute a vulnerable high-risk patient group and potentially benefit from targeted treatment.

Currently, the distribution of HPR- and LPR patients and their association with acute pain following UKA is not well investigated. The generated knowledge from this research project is essential to determine how studies with analgesia interventions should be designed. In the future, this will contribute to targeting treatment for high-risk patient groups to reduce pain and improve postoperative mobilization, and ultimately decrease the length of hospital stay in patients undergoing UKA. By targeting treatment, a potential overtreatment is also avoided.

Aim:

To investigate the prevalence of high- and low-pain responders, defined by a PCS score > 20 and ≤ 20 respectively, as well as the acute postoperative course of pain for these groups after unicompartmental knee arthroplasty.

Study location:

The inclusion will take place at the Dept. of Orthopaedic Surgery, Arthroplasty unit at Hvidovre Hospital, Capital Region of Denmark.

Study plan:

In the outpatient clinic, the screening procedure will be performed among patients planned to UKA by the surgeons. Patients will be asked if they may be contacted with the purpose of participating in a research project. Patients will undergo a preliminary examination where, as a standard procedure, the patient will receive a PCS questionnaire. Patients will be informed of the research project either in the outpatient clinic or by phone from an investigator.

All patients will receive verbal and written information about the project. All patients must give a signed informed consent on paper prior to inclusion to participate in the study.

Data protection:

All patient-related information will be treated confidentially, and data will be pseudoanonymized. Signed informed consent from participating patients will be stored at the Anesthesiologic Dept. 542, Hvidovre Hospital, in a locked cabinet. All electronic data will be stored in REDCap.

Collected variables:

During the hospital stay, data will be collected by contacting the patient at the Orthopaedic Dept. and by accessing the electronic patient journal. After discharge patients will be asked to fill out an electronic pain diary until 7 days after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral UKA
* Age ≥ 18 years
* Ability to participate in the study (understand written and spoken Danish language, self-reported pain and satisfaction).
* Filled out the Pain Catastrophizing Scale preoperatively.
* Signed written informed consent form.

Exclusion Criteria:

* Mental disability that could impair a patient's decision-making capability of giving informed consent and not enabling valid data collection.
* Insulin-treated diabetes mellitus
* Patients with known diagnoses of schizophrenia, ongoing psychosis, bipolar disease and/or a history of ongoing anti-psychotic treatment.
* Patients with modulated pain-reception (experience) based on other diseases or injuries, e.g. spinal cord or brain injury, severe polyneuropathies or neurologic disorders.
* Peripheral nerve block per- or postoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for unicompartmental knee arthroplasty at a Danish hospital.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Ratio between HPR:LPR patients defined as patients with PCS > 20 and PCS ≤ 20 respectively | Preoperatively

SECONDARY OUTCOMES:
Incidence of moderate to severe pain (VAS > 30 mm) during a 5-meter walk test 24 hours postoperatively in LPR patients | 24 hours
Incidence of moderate to severe pain (VAS > 30 mm) during a 5-meter walk test 24 hours postoperatively in HPR patients | 24 hours

OTHER OUTCOMES:
Difference between HPR:LPR patients in incidence of moderate to severe pain (VAS > 30 mm) during a 5-meter walk test 24 hours postoperatively | 24 hours
Difference between HPR:LPR patients in incidence of moderate to severe pain (VAS > 30 mm) at rest 24 hours postoperatively | 24 hours
Difference between HPR:LPR patients in cumulated pain upon ambulation in a 5-meter walk test day 2-7 | Day 2-7
Difference between HPR:LPR patients in cumulative use of rescue-analgesics per day in hospital day 0 to discharge, and at home from day of discharge to day 7 | Day 0-7
Difference between HPR:LPR patients in quality of sleep, lethargy, dizziness and nausea pre- and postoperatively from day 0 to day 7 | Day 0-7
Difference between HPR:LPR patients in length of stay | Day 0-7

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai B Foss, MD, dr.med., Study Director — Department of Anaesthesiology, Copenhagen University Hospital Hvidovre
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The individual patient data will be made available in anonymized form.
Supporting Information: SAP
Time Frame: Data will be available from the date of publication.

REFERENCES:
- [Background] Beard DJ, Davies LJ, Cook JA, MacLennan G, Price A, Kent S, Hudson J, Carr A, Leal J, Campbell H, Fitzpatrick R, Arden N, Murray D, Campbell MK; TOPKAT Study Group. The clinical and cost-effectiveness of total versus partial knee replacement in patients with medial compartment osteoarthritis (TOPKAT): 5-year outcomes of a randomised controlled trial. Lancet. 2019 Aug 31;394(10200):746-756. doi: 10.1016/S0140-6736(19)31281-4. Epub 2019 Jul 17. PMID 31326135
- [Background] Birch S, Stilling M, Mechlenburg I, Hansen TB. The association between pain catastrophizing, physical function and pain in a cohort of patients undergoing knee arthroplasty. BMC Musculoskelet Disord. 2019 Sep 12;20(1):421. doi: 10.1186/s12891-019-2787-6. PMID 31511076
- [Background] Hansen EN, Ong KL, Lau E, Kurtz SM, Lonner JH. Unicondylar Knee Arthroplasty Has Fewer Complications but Higher Revision Rates Than Total Knee Arthroplasty in a Study of Large United States Databases. J Arthroplasty. 2019 Aug;34(8):1617-1625. doi: 10.1016/j.arth.2019.04.004. Epub 2019 Apr 8. PMID 31064725
- [Background] Inacio MCS, Paxton EW, Graves SE, Namba RS, Nemes S. Projected increase in total knee arthroplasty in the United States - an alternative projection model. Osteoarthritis Cartilage. 2017 Nov;25(11):1797-1803. doi: 10.1016/j.joca.2017.07.022. Epub 2017 Aug 8. PMID 28801208
- [Background] Jensen CB, Petersen PB, Jorgensen CC, Kehlet H, Troelsen A, Gromov K; Lundbeck Foundation Centre for Fast-track Hip and Knee Replacement Collaborative Group. Length of Stay and 90-Day Readmission/Complication Rates in Unicompartmental Versus Total Knee Arthroplasty: A Propensity-Score-Matched Study of 10,494 Procedures Performed in a Fast-Track Setup. J Bone Joint Surg Am. 2021 Jun 16;103(12):1063-1071. doi: 10.2106/JBJS.20.01287. PMID 33784260
- [Background] Jensen CB, Troelsen A, Nielsen CS, Otte NKS, Husted H, Gromov K. Why are patients still in hospital after fast-track, unilateral unicompartmental knee arthroplasty. Acta Orthop. 2020 Aug;91(4):433-438. doi: 10.1080/17453674.2020.1751952. Epub 2020 Apr 14. PMID 32285727
- [Background] Kim MS, Koh IJ, Choi YJ, Lee JY, In Y. Differences in Patient-Reported Outcomes Between Unicompartmental and Total Knee Arthroplasties: A Propensity Score-Matched Analysis. J Arthroplasty. 2017 May;32(5):1453-1459. doi: 10.1016/j.arth.2016.11.034. Epub 2016 Nov 27. PMID 27979407
- [Background] Liddle AD, Pandit H, Judge A, Murray DW. Patient-reported outcomes after total and unicompartmental knee arthroplasty: a study of 14,076 matched patients from the National Joint Registry for England and Wales. Bone Joint J. 2015 Jun;97-B(6):793-801. doi: 10.1302/0301-620X.97B6.35155. PMID 26033059
- [Background] Lunn TH, Frokjaer VG, Hansen TB, Kristensen PW, Lind T, Kehlet H. Analgesic effect of perioperative escitalopram in high pain catastrophizing patients after total knee arthroplasty: a randomized, double-blind, placebo-controlled trial. Anesthesiology. 2015 Apr;122(4):884-94. doi: 10.1097/ALN.0000000000000597. PMID 25782644
- [Background] Lunn TH, Gaarn-Larsen L, Kehlet H. Prediction of postoperative pain by preoperative pain response to heat stimulation in total knee arthroplasty. Pain. 2013 Sep;154(9):1878-1885. doi: 10.1016/j.pain.2013.06.008. Epub 2013 Jun 12. PMID 23769717
- [Background] Nemes S, Rolfson O, W-Dahl A, Garellick G, Sundberg M, Karrholm J, Robertsson O. Historical view and future demand for knee arthroplasty in Sweden. Acta Orthop. 2015;86(4):426-31. doi: 10.3109/17453674.2015.1034608. Epub 2015 Mar 25. PMID 25806653
- [Background] Ode Q, Gaillard R, Batailler C, Herry Y, Neyret P, Servien E, Lustig S. Fewer complications after UKA than TKA in patients over 85 years of age: A case-control study. Orthop Traumatol Surg Res. 2018 Nov;104(7):955-959. doi: 10.1016/j.otsr.2018.02.015. Epub 2018 Apr 21. PMID 29684539
- [Background] Otero JE, Gholson JJ, Pugely AJ, Gao Y, Bedard NA, Callaghan JJ. Length of Hospitalization After Joint Arthroplasty: Does Early Discharge Affect Complications and Readmission Rates? J Arthroplasty. 2016 Dec;31(12):2714-2725. doi: 10.1016/j.arth.2016.07.026. Epub 2016 Aug 9. PMID 27600301
- [Background] Pavlin DJ, Sullivan MJ, Freund PR, Roesen K. Catastrophizing: a risk factor for postsurgical pain. Clin J Pain. 2005 Jan-Feb;21(1):83-90. doi: 10.1097/00002508-200501000-00010. PMID 15599135
- [Background] Pinto PR, McIntyre T, Ferrero R, Almeida A, Araujo-Soares V. Predictors of acute postsurgical pain and anxiety following primary total hip and knee arthroplasty. J Pain. 2013 May;14(5):502-15. doi: 10.1016/j.jpain.2012.12.020. Epub 2013 Mar 27. PMID 23541065
- [Background] Wilson HA, Middleton R, Abram SGF, Smith S, Alvand A, Jackson WF, Bottomley N, Hopewell S, Price AJ. Patient relevant outcomes of unicompartmental versus total knee replacement: systematic review and meta-analysis. BMJ. 2019 Feb 21;364:l352. doi: 10.1136/bmj.l352. PMID 30792179
- [Background] Nielsen NI, Kehlet H, Gromov K, Troelsen A, Husted H, Varnum C, Kjaersgaard-Andersen P, Rasmussen LE, Pleckaitiene L, Foss NB. High-dose steroids in high pain responders undergoing total knee arthroplasty: a randomised double-blind trial. Br J Anaesth. 2022 Jan;128(1):150-158. doi: 10.1016/j.bja.2021.10.001. Epub 2021 Nov 5. PMID 34749994

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT05510947/Prot_SAP_000.pdf